CLINICAL TRIAL: NCT07242638
Title: Use of Specific JAK Inhibition on Inflammatory Skin and Scalp Diseases in Down Syndrome R61AR084210
Brief Title: Treatment of Atopic Dermatitis and Alopecia Areata With Abrocitinib in Individuals With Down Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Columbia University (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Emma Guttman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-00773; 1R61AR084210 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Alopecia Areata
Keywords: Down Syndrome; Atopic Dermatitis; Alopecia Areata; Abrocitinib
MeSH Terms: conditions — Dermatitis, Atopic; Alopecia Areata; Down Syndrome | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Abrocitinib (Experimental): Participants with DS with either AD or AA will be given Abrocitinib 100mg. In the case where patients is not responsive to treatment at Week 12 per protocol defined non-responder criteria, the treatment dosage will change to Abrocitinib 200 mg.
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — All participants will be started on 100mg Abrocitinib daily. Based on clinical response, non-responders will be increased to 200mg daily at week 12. Responders will continue to receive 100 mg dose of Abrocitinib. All AA and AD participants will be maintained on their dose of Abrocitinib through week 60.

SUMMARY:
This is a single-center, open-label, basket phase 2b trial that will enroll Down Syndrome (DS) participants with at least one inflammatory skin condition (Atopic Dermatitis (AD) and/or Alopecia Areata (AA)). Patients will receive Abrocitinib 100 mg daily for 12 weeks. Responders (defined as achieving Eczema Area and Severity Index (EASI) 75 response for AD, or SALT <= 20 for AA) will be kept on this dose, and non-responders based on these definitions, will initiate 200 mg daily for another 12 weeks. All AD and AA patients will be maintained on the respective dose of Abrocitinib from Week 24 through week 60.

DETAILED DESCRIPTION:
This is a single-center, open-label, basket phase 2b trial that will enroll DS subjects with at least one inflammatory skin condition (Atopic Dermatitis [AD] and/or Alopecia Areata [AA]). As our goal is to have 51 patients complete the study, with an estimated dropout rate of ~10%, we will enroll a total of n=56 patients. Patients will receive abrocitinib 100 mg daily for 12 weeks. Responders (defined as achieving EASI75 response for AD, or SALT ≤20 for AA) will be kept on this dose, and non-responders based on these definitions, will initiate 200 mg daily for another 12 weeks. All AD and AA patients will be maintained on their respective dose of abrocitinib from Week 24 through week 60.

Patients with AD and AA will have clinical evaluations as well as skin and blood specimens collected for molecular analysis at multiple time points. For AD patients, lesional and non-lesional tape strips will be collected at weeks 0, 12, 24, 48 and 60, and processed as we previously published. For AA patients, optional 2mm biopsies will be collected from lesional and non-lesional scalp at baseline and from lesional scalp at weeks 24 and 48. Blood samples (a total of 17mL at each visit, with 12mL dedicated to mechanistic analyses), will be collected at weeks 0, 12, 24, 36, 48, and 60.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible as study participants:

* Male or female participants who are at least 12 years old, for whom signed informed consent can be provided by parent or legal guardian/LAR prior to participation in any study assessments or procedures.
* Diagnosis of Trisomy 21 or translocation Down Syndrome.
* Participant is able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Week 0/Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product (IP), FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below: a. Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; or b. Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]).
* Participant has a history of ≥6 months AD (≥7%BSA) or AA (≥25% scalp involvement). If the participant presents with both conditions, but only one meets the inclusion criteria, then the participant can only be enrolled under that category. If a participant meets inclusion criteria for both conditions at the Baseline visit, then the participant will be enrolled under the AA category as this disease is less prevalent. If the AA category has fulfilled its enrollment target, then the participant will be enrolled in the AD category.
* Participant is judged to be in otherwise good overall health following a detailed medical and medication history, physical examination, and laboratory testing.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for randomization as study participants:

* Inability or unwillingness of a participant's parent or legal guardian/LAR to give written informed consent or comply with study protocol.
* Participant is pregnant or breastfeeding.
* Participants with AA: A. cause of hair loss is indeterminable and/or they have concomitant causes of alopecia, such as traction, cicatricial, pregnancy-related, druginduced, telogen effluvium, or advanced androgenetic alopecia (i.e. Ludwig Type III or Norwood-Hamilton Stage ≥ V). B. Participant has a history of AA with no evidence of hair regrowth for ≥7 years since the last episode of hair loss
* Participant has increased risk of developing venous thromboembolism, e.g. deep vein thrombosis or pulmonary embolism (history of venous thromboembolism, or first-degree relative with unprovoked venous thromboembolism (i.e. without known underlying cause such as trauma, surgery, immobilization, prolonged travel, pregnancy, hormone use, or plaster cast), that would suggest participant is at increased risk of inherited coagulation disorder (e.g. Factor V Leiden).
* Participant currently has active forms of other inflammatory skin diseases (eg, psoriasis, seborrheic dermatitis, lupus) at the time of Day 1 that would interfere with evaluation of AD or AA.
* Participant was vaccinated or exposed to a live or attenuated vaccine within the 6 weeks prior to Baseline visit, or is expected to be vaccinated or to have household exposure to these vaccines during treatment.
* Participant has a suspected or active lymphoproliferative disorder or malignancy; OR a history of malignancy within 5 years before the Week 0/Baseline assessment, except for completely treated in situ non-melanoma skin and cervical cancers without evidence of metastasis.
* Infection History: • Participant has an active bacterial, viral, or helminth parasitic infection; OR a history of ongoing, recurrent severe infections requiring systemic antibiotics. • Participant has active chronic or acute skin infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to Baseline or superficial skin infections within 1 week prior to Baseline. • Participant has a history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
* Participant has a history of alcohol or substance abuse within 6 months prior to Day 1 that in the opinion of the investigator will preclude participation in the study.
* Participant with a known or suspected underlying immunodeficiency or immune-compromised state as determined by the investigator.
* Participant has a concurrent or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, intestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease. ANY of the following abnormalities in renal or hepatic tests at screening are exclusionary: Estimated creatinine clearance <40 mL/min based on the age appropriate calculation, or serum creatinine >1.5 times the upper limit of normal (ULN); • Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >2 times the ULN; • Total bilirubin ≥1.5 times the ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN.
* Participant has active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) prior to Baseline.
* Participant has positive or indeterminable PPD or QFT result including participants that completed standard tuberculosis therapy prior to Baseline.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
* Participant has history of adverse systemic or allergic reactions to any component of the study drug or any safety event deemed "related" to a JAK inhibitor.
* Participant has used systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, oral JAK inhibitor (tofacitinib, ruxolitinib, baricitinib, ritlecitinib, or investigational oral JAK Inhibitors) or ultraviolet (UV) phototherapy with/without Psoralen Ultraviolet A (PUVA) therapy, within 4 weeks prior to the Week 0/Baseline visit.
* Participant has used systemic monoclonal antibody treatments (such as the IL-4R antagonist dupilumab) within 12 weeks of Baseline visit.
* Participant has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus within 1 week prior to the Week 0/Baseline visit.
* Participant with Translocation or Mosaic Downs Syndrome.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events (SAEs) at Week 24 and Week 60 | Week 24 and Week 60
  Rate of Serious Adverse Events (SAEs) at week 24 and at 60 weeks to assesses the clinical safety of Abrocitinib in patients with DS and AD or AA.

SECONDARY OUTCOMES:
Number and Severity of SAEs and TEAEs at Weeks 4, 8, 12 | Weeks 4, 8, 12
  Overall number and severity of SAEs and Treatment-Emergent Adverse Events (TEAEs) at weeks 4, 8, and 12.
Number of SAEs and TEAEs | Weeks 16, 28, 36, 48, 60
  Number and severity of SAEs and Treatment-Emergent Adverse Events (TEAEs) at weeks 16, 28, 36, 48 and 60 in each dose group
Proportion of Participants with AD Reaching EASI 75 | Week 24
  The proportion of subjects with AD achieving EASI 75 at week 24. The proportion of patients who achieve an improvement of 75% or greater at week 24. The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
Proportion of Participants with AA reaching SALT ≤ 20 | Week 24
  The proportion of subjects with AA achieving SALT ≤ 20 at week 24. SALT ≤ 20 is defined as the proportion of patients achieving ≤ 20% reduction in SALT score compared to baseline.
  Scalp is divided into 4 areas namely, Vertex - 40% (0.4) of scalp surface area; right profile of scalp - 18% (0.18) of scalp surface area; left profile of scalp - 18% (0.18) of scalp surface area; Posterior aspect of scalp - 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is percentage hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all above mentioned areas.
Change in proportions of participants with AD from baseline to Week 60 | Baseline to Week 60
  Change in proportions of patients achieving EASI 75 in participants with AD from baseline to week 60.
  The change in proportion of patients who achieve an improvement of 75% or greater from their Baseline EASI score to week 60. The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
Change in Proportion of AA participants with SALT <=20 at Week 60 | Baseline and Week 60
  Change in proportion of AA patients with SALT ≤20 at week 60 compared to baseline in each treatment and dose group.
  SALT ≤ 20 is defined as the proportion of patients achieving ≤ 20% reduction in SALT score compared to baseline.
  Scalp is divided into 4 areas namely, Vertex - 40% (0.4) of scalp surface area; right profile of scalp - 18% (0.18) of scalp surface area; left profile of scalp - 18% (0.18) of scalp surface area; Posterior aspect of scalp - 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is percentage hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all above mentioned areas.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Dusan Bogunovic, PhD, Principal Investigator — Columbia University
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be analyzed and published as aggregate data